CLINICAL TRIAL: NCT05744765
Title: Short And Long Term Effects Of Breathing Exercises on Reaction Time: A Randomized Controlled Trial
Brief Title: Effects of Breathing Exercises on Reaction Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Burçin Akçay, Assistant professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Bandırma Onyedi EylulU
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Breathing, Mouth
MeSH Terms: conditions — Mouth Breathing | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Randomized controlled, single-blind
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing exercises (Experimental): First evaluation - breathing exercises (1 session) - second evaluation - breathing exercises (11 sessions) - third evaluation
  Interventions: Other: breathing exercises
- No exercise (No Intervention): First evaluation - no intervention (1 session) - second evaluation - no intervention (11 sessions) - third evaluation

INTERVENTIONS:
Other: breathing exercises — After the initial 5 minutes of relaxed breathing, the participants will perform diaphragmatic and costal breathing for 10 minutes. .5 diaphragmatic breathing will be done in 1 minute.
  Arms: Breathing exercises

SUMMARY:
The aim of the study was to investigate the short and long-term effects of breathing exercises on reaction time.

DETAILED DESCRIPTION:
A total of 40 participants who volunteered to participate in the study from the students of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Bandırma Onyedi Eylül University will be included in the study. Participants will be randomly divided into two groups using a simple random numbers table. The study group (15 people) will be given respiratory exercises (12 sessions). The control group (15 people) will receive no intervention. In the study, after the demographic characteristics of the participants are obtained, reaction time will be evaluated with auditory and visual reaction tests and upper extremity reaction tests. All evaluations are planned to take a total of 15 minutes.

The same assessments will be performed in both groups. To measure the long-term effect, after the initial evaluations are completed, the study group will be given a total of 12 sessions of breathing exercises for 4 weeks (3 days a week). After 4 weeks, both groups will be evaluated again. To measure the short-term effect, the respiratory exercise program will be started after the 1st evaluation in the study group, and the 2nd evaluation will be made after the first session.

Canan Demir will perform breathing exercises, and the other researchers who will evaluate will not know which group the participants are in. In this way, the study will be single-blinded.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* To be between the ages of 18-30
* Not having any problems that prevent breathing exercises

Exclusion Criteria:

* Acute infection or chronic disease of neurological, psychiatric, orthopedic, cardiological, rheumatological, etc. origin
* Having had any injury and/or operation (trauma, surgery, fracture, etc.) in the last 6 months
* Regular medication use
* Presence of respiratory disease (asthma, COPD, etc...)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Finger reaction test | 4weeks
  By placing the dominant hand index finger on the left button of a computer mouse, the participant will be asked to press the left button as soon as the traffic light pattern glows green on the screen.
Upper extremity reaction test | 4weeks
  Upper extremity reaction test: It is planned to use a validated BlazePod sensor for upper extremity reaction time test
Auditory Reaction Test | 4weeks
  Auditory reaction time will be assessed with the playback.fm (https://playback.fm/audio-reaksiyon-time) test. Subjects will be asked to press the 'space bar' key each time they hear a sound. After five applications, data will be taken from the output page and the average reaction time will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- BandırmaOnyediEylulU, Balıkesir, Turkey (Türkiye)